CLINICAL TRIAL: NCT00593684
Title: The Safety Evaluation of Silver Alginate (Algidex™) Dressing in Very Low Birth Weight (VLBW) Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: DeRoyal Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 005-206; 0000
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Prematurity; Very Low Birth Weight
Keywords: neonate; central lines; very low birth weight; silver alginate
MeSH Terms: conditions — Premature Birth

ARMS (2):
- Algidex patch (Experimental): Infants in this group received the Algidex patch on top of the line insertion sites of any of the following lines: umbilical arterial line, umbilical venous line, peripheral arterial line, peripheral long line, and central venous line. This is a sterile patch of polyurethane foam coated with silver alginate and maltodextrin matrix that is impregnated with 141 mg of ionic silver per 100 cm2. Every 7 days, each insertion site was cleansed and then a new patch was placed and covered with a fresh occlusive dressing (Tegaderm, Opsite).
  Interventions: Device: Silver Alginate
- Control group (No Intervention): Infants in this group served as the control group and received line-dressing changes every 7 days according to standard hospital protocol specific for the type of line inserted. Insertion sites were covered with only an occlusive dressing (Tegaderm, Opsite).

INTERVENTIONS:
Device: Silver Alginate — This is a sterile patch of polyurethane foam coated with silver alginate and maltodextrin matrix that is impregnated with 141 mg of ionic silver per 100 cm2.
  Other Names: Algidex™ extra small patches
  Arms: Algidex patch

SUMMARY:
The purpose of this study is to test the safety of silver alginate (Algidex™) dressing in VLBW infants in preparation for a large efficacy trial.

DETAILED DESCRIPTION:
We are conducting a pilot randomized controlled trial in VLBW infants to evaluate the safety of silver alginate (Algidex™) dressing compared to standard catheter care. Following parental consent, infants are randomized to receive silver alginate or standard of care dressing. Infants with birth weights less than 1,500 grams admitted to Baylor University Medical Center (BUMC) NICU with any of the following lines are eligible for inclusion into this study up to 72 hours after birth: umbilical arterial line (UAL), umbilical venous line (UVL), peripheral arterial line (PAL), peripheral long line (PLL), and central venous line (CVL). Safety is assessed by measuring silver levels and monitoring for cutaneous reactions. Dressings are changed every seven days. Silver levels are drawn on study days 1, 7, and 28. Blood culture results are used to compare infection rates between the two groups. Patient demographics and clinical conditions are recorded. Results will be analyzed based on intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weights less than 1,500 grams admitted to Baylor University Medical Center (BUMC) NICU with any of the following lines are eligible for inclusion into this study up to 72 hours after birth: umbilical arterial line (UAL), umbilical venous line (UVL), peripheral arterial line (PAL), peripheral long line (PLL), and central venous line (CVL).

Exclusion Criteria:

* N/A

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Furgan Moin, M.D., Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center - Women and Children's Services, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at the Baylor University Medical Center Neonatal Intensive Care Unit between April 2006 and December 2007.
Pre-assignment Details: Enrollment and group assignment occurred concurrently.
Groups:
- Control: Infants in this group served as the control group and received line-dressing changes every 7 days according to standard hospital protocol specific for the type of line inserted. Insertion sites were covered with only an occlusive dressing (Tegaderm, Opsite).
Period: Overall Study
Arm/Group | Algidex Patch | Control
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Algidex Patch | Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: weeks] — weeks of gestation
  weeks | 27.3 (2.03) | 27.2 (1.85) | 27.25 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 3 | 15 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11
Birth Weight (grams) [Mean (Standard Deviation); unit: Grams] | 955 (250) | 913 (209) | 934 (229)
Average Line Days [Mean (Standard Deviation); unit: line days] — umbilical arterial line, umbilical venous line, peripheral arterial line, peripheral long line, and central venous line calculated per 1,000 days.
  line days | 17.95 (8.8) | 19 (9.9) | 18.5 (9.35)

OUTCOME MEASURES:

1. Primary Outcome: Serum Silver Concentration at 1 Day
Description: Serum silver concentrations were obtained from both groups on study days 1, 7, and 28. Study day 1 was defined as the 24 hour period in which participants enrolled in the study. Here we are examining the results of first day, or 24 hours from enrollment. Silver samples were analyzed using a dual inductively coupled plasma -mass spectrometry methodology. Accepted reference values for non-exposure silver concentrations are defined as <15 ng ml -1 with standard Mayo Clinic reference technique.
Time Frame: 1 Day (first 24 hours from enrollment)
Population: Study design included intent-to-treat for data collection and intention to stop if signs of toxicities or adverse effects were noted.
Measure: Mean (Standard Deviation); unit: ng ml -1
Groups:
- Algidex Patch: The group of patients that were randomized to receive the Algidex patch during the study.
Arm/Group | Algidex Patch | Control
Number analyzed (Participants) | 25 | 24
ng ml -1 | 7.6 (20.93) | 0.22 (0.09)

2. Primary Outcome: Serum Silver Concentration at 7 Days
Description: Serum silver concentrations were obtained from both groups on study days 1, 7, and 28. Study day 1 was defined as the 24 hour period in which participants enrolled in the study. Here we examine the results at 7 days from enrollment. Silver samples were analyzed using a dual inductively coupled plasma -mass spectrometry methodology. Accepted reference values for non-exposure silver concentrations are defined as <15 ng ml -1 with standard Mayo Clinic reference technique.
Time Frame: 7 Days from enrollment
Population: One subject in each group died
Measure: Mean (Standard Deviation); unit: ng ml -1
Arm/Group | Algidex Patch | Control
Number analyzed (Participants) | 24 | 24
ng ml -1 | 4.79 (4.37) | 0.23 (0.14)

3. Primary Outcome: Serum Silver Concentrate at 28 Days
Description: Serum silver concentrations were obtained from both groups on study days 1, 7, and 28. Study day 1 was defined as the 24 hour period in which participants enrolled in the study. Here we examine results at 28 days from enrollment. Silver samples were analyzed using a dual inductively coupled plasma -mass spectrometry methodology. Accepted reference values for non-exposure silver concentrations are defined as <15 ng ml -1 with standard Mayo Clinic reference technique.
Time Frame: 28 Days from enrollment
Population: two subjects died in the treatment group; one subject died in the control group
Measure: Mean (Standard Deviation); unit: ng ml -1
Arm/Group | Algidex Patch | Control
Number analyzed (Participants) | 23 | 24
ng ml -1 | 3.19 (3.23) | 0.21 (0.07)

4. Secondary Outcome: Infection Rate
Description: Infection was defined as recovery of a bacterial pathogen or fungus from any single blood culture. Infection rate was defined as Infections/1000 line days.
Time Frame: infection per 1,000 Line Days
Measure: Number; unit: Infection per 1,000 line days
Arm/Group | Algidex Patch | Control
Number analyzed (Participants) | 25 | 24
Infection per 1,000 line days | 6.69 | 12.34

ADVERSE EVENTS:
Time Frame: Time of enrollment (signed consent) until hospital discharge.
Description: Serum Silver concentration measures ended at day 28 and/or when central line discontinued
Arm/Group | Algidex Patch | Control
Serious Adverse Events (participants affected / at risk) | 2/25 | 4/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Algidex Patch (N=25) | Control (N=25)
Death (Pregnancy, puerperium and perinatal conditions) | 2 | 4 — Complications of prematurity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes